CLINICAL TRIAL: NCT07018869
Title: A Pragmatic Randomized Controlled Trial to Evaluate the Effectiveness of an Intervention Called Current Together After Cancer (CTAC) to Promote Guideline-Concordant Colorectal Cancer Surveillance
Brief Title: Evaluating Whether an Educational Website Called Current Together After Cancer (CTAC) Improves Follow-up Care for Colorectal Cancer Survivors
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: S2417CD; NCI-2025-03080 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2417CD (Other: SWOG); SWOG-S2417CD (Other: DCP); S2417CD (Other: CTEP); R01CA293394 (NIH); UG1CA189974 (NIH)
Record Dates: First submitted 2025-05-21; First posted 2025-06-13 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer Stage II; Colorectal Cancer Stage III
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (CTAC) (Experimental): Patients and supporter participants receive access to the CTAC intervention website and may review the content as frequently as they like for up to 16 months on study.
  Interventions: Other: Intervention website access; Other: Interview; Other: Questionnaire Administration
- Group 2 (Control) (Active Comparator): Patients and supporter participants receive access to a general health education website and may review the content as frequently as they like for up to 16 months on study.
  Interventions: Other: Control website access; Other: Interview; Other: Questionnaire Administration

INTERVENTIONS:
Other: Intervention website access — Receive access to CTAC intervention website with educational content and interactive modules
  Arms: Group 1 (CTAC)
Other: Control website access — Receive access to CTAC control website with general health education
  Arms: Group 2 (Control)
Other: Interview — Ancillary studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial evaluates whether a web-based intervention called Current Together after Cancer (CTAC) works to increase the number of patients with surgically removed (resected) colorectal cancer who receive surveillance care that aligns with current guidelines (guideline-concordant). Surveillance care after resection of colorectal cancer is critical to detect potentially curable return of disease (recurrence), yet up to 60% of colorectal cancer survivors fail to receive surveillance. This may be due to a lack of knowledge about the purpose of surveillance care and the risks of cancer recurrence, or a lack of confidence for managing surveillance care. The CTAC intervention is an online education intervention designed to improve patients' knowledge about surveillance and their self-efficacy for managing surveillance, and to promote effective communication with supporters and supporter engagement in patients' surveillance in a way that is aligned with each patient's preferences. By increasing a patient's knowledge, self-efficacy, and satisfaction with their supporter's engagement in their care, the CTAC intervention may increase the number of patients who receive guideline-concordant surveillance care after resection of colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate whether the patients randomized to the Current Together After Cancer (CTAC) intervention website compared to the CTAC control website have higher rates of guideline-concordant colorectal cancer (CRC) surveillance at 12 months after registration.

SECONDARY OBJECTIVES:

I. To assess patient reported knowledge about surveillance at 3 and 16 months post-patient registration. (Comparing CTAC intervention versus [vs.] control) II. To assess patient reported self-efficacy in management of surveillance 3 and 16 months post-patient registration using previously developed CRC screening self-efficacy measure. (Comparing CTAC intervention vs. control) III. To assess patient reported satisfaction with supporter engagement in surveillance 3 and 16 months post-patient registration. (Comparing CTAC intervention vs. control)

EXPLORATORY OBJECTIVES:

I. To assess the implementation of CTAC into clinic workflow, and to better understand barriers and facilitators to the delivery of the intervention arm using a mixed-methods approach. (For the process evaluation of the CTAC intervention) II. To explore the association between supporter participation in the assigned CTAC intervention at 3 months with receipt of CRC surveillance at 16 months. (Regarding supporter participation) III. To explore the association between supporter participation in the assigned CTAC intervention at 3 months with knowledge about surveillance; at 16 months. (Regarding supporter participation) IV. To explore the association of supporter participation in the assigned CTAC intervention at 3 months with self-efficacy in management of surveillance at 16 months. (Regarding supporter participation) V. To explore the association of supporter participation in the assigned CTAC intervention at 3 months. (Regarding supporter participation)

OUTLINE: Patients are randomized to 1 of 2 groups and supporter participants are assigned to the arm to which their patient was randomized.

GROUP 1: Patients and supporter participants receive access to the CTAC intervention website and may review the content as frequently as they like for up to 16 months on study.

GROUP 2: Patients and supporter participants receive access to a general health education website and may review the content as frequently as they like for up to 16 months on study.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS:
* Patient participants must have newly diagnosed surgically resected, stage II or stage III colorectal cancer per the timing described below
* Patient participants must have an adult in their life who supports them in their colorectal cancer journey who they might be willing to invite to join them in viewing an educational website. This is determined via the question: "Do you have an adult in your life, such as a spouse/partner, family member or friend, who supports you with your colorectal cancer journey and may be willing to view a website with you? When we say, "supports you in your colorectal cancer journey", we mean things like, helping you keep and get to medical appointments, talking with you and/or your doctors about your cancer, or helping you make decisions about your cancer."

  * Those who respond "no" to the question above will be told that "Because this study is for patients and a supporter to view the website together, you are not eligible for this study, but there may be other studies you are eligible for in the future".
  * NOTE: The above question will be used to define "supporter" for purposes of this study. Examples of supporters include a spouse, partner, sibling, adult child, another family member, or friend.
  * NOTE: The supporter does not have to agree to participate in the study in order for the patient to be eligible for this study. Justification for requiring the enrolled patient to have a supporter (whether the supporter is invited or participates) is based on the study's underlying conceptual framework
* Patient participants must not have recurrent or metastatic (stage IV) colorectal cancer
* Patient participants must not have a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the efficacy assessment of this intervention
* Patient participants must be registered within 90 - 180 days of surgical resection
* Patient participants must be ≥ 18 years of age at the time of registration/randomization. The lower cutoff of 18 was determined because the lower age range of patients that may be recruited to Southwest Oncology Group (SWOG) studies is 18
* Patient participants must have Zubrod performance status of 0-2
* Patient participants must be able to read English or Spanish since the website for the intervention and control arm are available in English and Spanish
* Patient participants must: 1) be able to complete Patient Reported Outcome (PRO) questionnaires in English or Spanish, and 2) agree to complete PROs at all scheduled timepoints
* Patient participants will be encouraged to provide an email address or cell phone number, if possible, for the purpose of being contacted by staff at the University of Michigan who will provide access to the educational website. For those who do not wish to provide or create an email address or a cell phone number, they may still participate with alternate methods
* Patient participants must not be enrolled or be planning to enroll in a clinical trial of investigational treatment that includes imaging and/or laboratory monitoring for the duration of this trial

  * NOTE: Patient participants are allowed to be co-enrolled on other non-treatment clinical trials
* SUPPORTER PARTICIPANT:
* Supporter participants must be ≥ 18 years of age at the time of registration/randomization
* Supporter participants must be able to read English or Spanish since the educational website is available in English and Spanish
* Supporter participants must have been identified by the patient as a person who may be willing to join them in reviewing the educational website
* PATIENT AND SUPPORTER:
* NOTE: As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

  * Patient and supporter participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines. This protocol does not permit use of Legally Authorized Representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1057 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2029-05-23 (Estimated); Study Completion 2029-06-06 (Estimated)

PRIMARY OUTCOMES:
Receipt of colorectal cancer surveillance | At 16 months
  Receipt of the four surveillance components will be abstracted as a binary outcome (yes versus no) from the electronic medical record for every enrolled patient. Additionally, patient-reported receipt of surveillance will be collected via survey. Multivariable logistic regression will be used, adjusted for the stratification factors as covariates.

SECONDARY OUTCOMES:
Knowledge About Colorectal Follow-Up Care score | At baseline, 3 months, and 16 months
  The Knowledge About Colorectal Follow-Up Care score is patterned after instruments used in prior research that measure knowledge about colorectal cancer screening. 5 questions are asked of participants about the purpose of colorectal cancer surveillance, what is included in surveillance, recommended timeframe for surveillance, recurrence, and odds of new colorectal cancer diagnosis compared to the general population. Each question will receive one point for a correct answer and 0 points for an incorrect answer. One question is written as "select all that apply"; all correct answers must be selected for the question to count as correctly answered. The number of correct answers will be summed to give an overall knowledge score (ranging from 0 to 5). Change in knowledge over time will be compared between the two arms using multivariable logistic regression. Regression models will adjust for the stratification variables as covariates.
Cancer Worry Scale (CWS) | At baseline, 3 months, and 16 months
  8-item scale detecting fear of recurrence in cancer survivors, rated on a 4-item Likert scale ranging from "never" to "almost always." Scores range from 8 to 32, with a higher total score indicating greater worry about cancer and/or greater impact on mood and daily functioning. Multivariable logistic regression will be used. Regression models will adjust for the stratification variables as covariates.
Follow-up care preferences questionnaire | At baseline, 3 months, and 16 months
  The follow-up care preferences questionnaire is a 9-item questionnaire that solicits participants' preferences about follow-up care (i.e., "When thinking about your colorectal cancer follow-up care, how important to you are the following?") with questions (e.g., "It keeps you from worrying about the cancer coming back") answered using a 5-item Likert scale ranging from "Not at all important" to "Very important." Changes in preferences over time will be described and reported by arm.
Self-efficacy for managing follow-up care | At baseline, 3 months, and 16 months
  This scale is adapted with permission from a 6-item scale used to measure colorectal cancer screening self-efficacy. Responses to individual questions are scored from 1 to 5 with higher values representing higher self-efficacy. An overall score is calculated by averaging the individual question scores. Multivariable linear regression will be used for analysis. Regression models will adjust for the stratification variables as covariates.
Patient Reported Outcomes Measurement Information System (PROMIS)-29 + 2 Profile version 2.1, Physical Function Measure only | At baseline, 3 months, and 16 months
  Physical Function (PF) Measure taken from PROMIS-29+2 Profile version 2.1. 4 questions measuring ability to perform standard physical daily tasks. Individual questions are rated on Likert scale from "Unable to do" to "Without any difficulty." Scores are generally converted to T-Scores, with a mean of 50 and a standard deviation of 10 in the general population. Higher scores represent better physical function. Multivariable linear regression will be performed with stratification factors included as covariates.
Satisfaction with supporter engagement questionnaire | At 3 months, and 16 months
  The satisfaction with supporter engagement questionnaire consists of two parts: questions measuring overall satisfaction with the supporter's involvement in the participant's colorectal cancer follow-up care (4 items, each rated on a 5-level Likert scale; completed at 3 months and 16 months) and one question asking about whether the participant chose to invite a supporter and whether the participant and supporter viewed their assigned website together (this question completed only at the 3-month timepoint).
  Each question will be reported and analyzed separately with multivariate linear regression using stratification factors as covariates.

OTHER OUTCOMES:
Barriers and facilitators of intervention uptake and use | Up to 16 months
  The analysis plan involves reviewing the audio recorded interviews and developing a coding scheme under each component of the Consolidated Framework for Implementation Research domains. This scheme will then be shared with the rest of the study team for review and discussion to pull out high level "themes" regarding barriers and facilitators of intervention uptake and use. These themes will be reported on in a subsequent usability manuscript.
Supporter participation/inclusion in the assigned intervention | Up to 16 months
  Will evaluate the association between supporter participation in the assigned intervention (evaluated at 3 months) and the following patient outcomes (evaluated at 16 months): 1) patient receipt of CRC surveillance, 2) patient knowledge about surveillance, 3) patient self-efficacy in management of surveillance, and 4) patient satisfaction with supporter engagement. Supporter inclusion in the assigned intervention at 3 months will be determined from responses to the Satisfaction with Supporter Engagement questionnaire. Analyses will be conducted using multivariable logistic regression.

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Veenstra, Principal Investigator — SWOG Cancer Research Network
Locations (341):
- United States (334):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Mercy Cancer Center, Merced, California
  - Providence Queen of The Valley, Napa, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Providence Medical Foundation - Santa Rosa, Santa Rosa, California
  - Providence Santa Rosa Memorial Hospital, Santa Rosa, California
  - Saint Joseph's Medical Center, Stockton, California
  - Woodland Memorial Hospital, Woodland, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Saint Anthony North Hospital, Westminster, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Augusta University Medical Center, Augusta, Georgia
  - Northeast Georgia Medical Center Braselton, Braselton, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - UI Healthcare Mission Cancer and Blood - Pella, Pella, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - The Iowa Clinic PC, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - MaineHealth Waldo Hospital, Belfast, Maine
  - MaineHealth Cancer Care and IV Therapy - Brunswick, Brunswick, Maine
  - MaineHealth LincolnHealth Hospital, Damariscotta, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth Cancer Care and IV Therapy - Sanford, Sanford, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - Christiana Care - Union Hospital, Elkton, Maryland
  - MyMichigan Medical Center Gratiot, Alma, Michigan
  - MyMichigan Medical Center Alpena, Alpena, Michigan
  - Trinity Health IHA - Obstetrics and Gynecology West Arbor, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - MyMichigan Medical Center Gladwin, Gladwin, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - MyMichigan Medical Center Mount Pleasant, Mount Pleasant, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Essentia Health - Baxter Clinic, Baxter, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Saint Joseph's Crosslake Clinic, Crosslake, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health - Ely Clinic, Ely, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health - International Falls Clinic, International Falls, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Essentia Health - Moose Lake Clinic, Moose Lake, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Essentia Health - Saint Joseph's Pequot Lakes Clinic, Pequot Lakes, Minnesota
  - Essentia Health - Saint Joseph's Pine River Clinic, Pine River, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Essentia Health - Saint Joseph's Staples Clinic, Staples, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Hi-Line Sletten Cancer Center, Havre, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Hood River Memorial Hospital, Hood River, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Sovah Health Martinsville, Martinsville, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Cancer Care Northwest-Valley, Spokane, Washington
  - Cancer Care Northwest-North Spokane, Spokane, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Essentia Health-Hayward Clinic, Hayward, Wisconsin
  - Tamarack Health Hayward Medical Center, Hayward, Wisconsin
  - ThedaCare Regional Medical Center - Neenah, Neenah, Wisconsin
  - ThedaCare Cancer Care - New London, New London, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - ThedaCare Cancer Care - Oshkosh, Oshkosh, Wisconsin
  - ThedaCare Cancer Care - Shawano, Shawano, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Sheboygan Physicians Group, Sheboygan, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - ThedaCare Cancer Care - Waupaca, Waupaca, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
- Puerto Rico (7):
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Puerto Rico Hematology Oncology Group, Bayamón
  - Doctors Cancer Center, Manatí
  - San Juan Community Oncology Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - PROncology, San Juan
  - San Juan City Hospital, San Juan